CLINICAL TRIAL: NCT00681213
Title: Tacrolimus and Mycophenolate Versus Tacrolimus and Sirolimus vs. Neoral and Sirolimus Used in Combination in Cadaver and Non-HLA Identical Living Related Kidney Transplants
Brief Title: Tacrolimus/Sirolimus Versus Tacrolimus/Mycophenolate Mofetil (MMF) Versus Neoral/Sirolimus in Adult, Primary Kidney Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Wyeth-Ayesrst Pharmaceuticals, Roche Laboratories, and Fujusawa Healthcare, Inc. (Unknown)
Responsible Party: Dr. George W. Burke, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB#19990664
Record Dates: First submitted 2008-05-19; First posted 2008-05-21 (Estimated); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Adult Primary Kidney Transplantation
MeSH Terms: interventions — Tacrolimus; Sirolimus; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Experimental): Tacrolimus/Sirolimus
  Interventions: Drug: Tacrolimus/Sirolimus
- B (Experimental): Tacrolimus/MMF
  Interventions: Drug: Tacrolimus/MMF
- C (Experimental): Neoral/Sirolimus
  Interventions: Drug: Neoral/Sirolimus

INTERVENTIONS:
Drug: Tacrolimus/Sirolimus
  Arms: A
Drug: Tacrolimus/MMF
  Arms: B
Drug: Neoral/Sirolimus
  Arms: C

SUMMARY:
Comparison of outcomes/safety/and tolerability of SRL/FK/Pred vs. FK/MMF/Pred vs. SRL/Neoral®/Pred in cadaveric and non-HLA identical LRD kidney transplants.

ELIGIBILITY:
Inclusion Criteria:

* Age >14 years
* Weight > 40 kg
* Primary renal allograft: cadaveric or mismatched living donor
* Negative standard cross match for T-cells
* Women of childbearing potential will be required to have a negative qualitative serum pregnancy test and agree to use an adequate method of contraception throughout the study period and for 3 months after discontinuation of study medication (3yrs, 3 mos.)
* Signed and dated informed consent (Parent or legal guardian must provide written consent for patients <18 years of age)

Exclusion Criteria:

* Evidence of systemic infection
* History of malignancy within 10 years (with the exception of localized skin cancer)
* Use of any investigational drug or treatment up to 4 weeks prior to enrolling in the study and during the 12-month treatment phase
* Concurrent use of astemizole, pimozide, cisapride, terfenadine, or ketoconazole
* Known hypersensitivity to sirolimus and its derivatives
* Patients with a screening/baseline (or within 96 hours of transplant)

  * total white blood cell count < 4000/mm3;
  * platelet count < 100,000/mm3;
  * fasting triglycerides > 400 mg/dl (> 4.6 mmol/L);
  * fasting total cholesterol > 300 mg/dl (> 7.8 mmol/L);
  * fasting HDL-cholesterol < 30 mg/dl;
  * fasting LDL-cholesterol > 200mg/dl

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2000-05; Primary Completion 2001-12 (Actual); Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of acute rejection episodes | 1 year

SECONDARY OUTCOMES:
1. Graft loss 2. Renal function as determined by serum creatinine and calculated creatinine clearance (using the Cockcroft-Gault method) six and 12 months | 1, 3, and 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- University of Miami Division of Transplantation, Miami, Florida, United States

REFERENCES:
- [Result] Ciancio G, Burke GW, Gaynor JJ, Mattiazzi A, Roth D, Kupin W, Nicolas M, Ruiz P, Rosen A, Miller J. A randomized long-term trial of tacrolimus and sirolimus versus tacrolimus and mycophenolate mofetil versus cyclosporine (NEORAL) and sirolimus in renal transplantation. I. Drug interactions and rejection at one year. Transplantation. 2004 Jan 27;77(2):244-51. doi: 10.1097/01.TP.0000101290.20629.DC. PMID 14742989
- [Result] Ciancio G, Burke GW, Gaynor JJ, Mattiazzi A, Roth D, Kupin W, Nicolas M, Ruiz P, Rosen A, Miller J. A randomized long-term trial of tacrolimus/sirolimus versus tacrolimus/mycophenolate mofetil versus cyclosporine (NEORAL)/sirolimus in renal transplantation. II. Survival, function, and protocol compliance at 1 year. Transplantation. 2004 Jan 27;77(2):252-8. doi: 10.1097/01.TP.0000101495.22734.07. PMID 14742990
- [Result] Ciancio G, Burke GW, Gaynor JJ, Ruiz P, Roth D, Kupin W, Rosen A, Miller J. A randomized long-term trial of tacrolimus/sirolimus versus tacrolimums/mycophenolate versus cyclosporine/sirolimus in renal transplantation: three-year analysis. Transplantation. 2006 Mar 27;81(6):845-52. doi: 10.1097/01.tp.0000203894.53714.27. PMID 16570006
- [Derived] Oliveras L, Lopez-Vargas P, Melilli E, Codina S, Royuela A, Coloma Lopez A, Fava A, Manonelles A, Couceiro C, Lloberas N, Cruzado JM, Montero N. Delayed initiation or reduced initial dose of calcineurin-inhibitors for kidney transplant recipients at high risk of delayed graft function. Cochrane Database Syst Rev. 2025 Apr 8;4(4):CD014855. doi: 10.1002/14651858.CD014855.pub2. PMID 40197799
- [Derived] Ciancio G, Gaynor JJ, Sageshima J, Roth D, Kupin W, Guerra G, Tueros L, Zarak A, Hanson L, Ganz S, Chen L, Ruiz P, Livingstone AS, Burke GW 3rd. Machine perfusion following static cold storage preservation in kidney transplantation: donor-matched pair analysis of the prognostic impact of longer pump time. Transpl Int. 2012 Jan;25(1):34-40. doi: 10.1111/j.1432-2277.2011.01364.x. Epub 2011 Oct 8. PMID 21981661